CLINICAL TRIAL: NCT00542919
Title: A Multicenter, Open-label, Noncomparative Study of Enzastaurin in Patients With Non-Hodgkin's Lymphomas
Brief Title: A Study for Patients With Non-Hodgkin's Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11503; H6Q-MC-S057 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: T-Cell Lymphoma; B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, B-Cell | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- T-Cell (Experimental): T-Cell (TCL): Peripheral and cutaneous T-cell lymphoma (PTCL, CTCL). Participants received enzastaurin 1125 milligram (mg) loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days
  Interventions: Drug: enzastaurin
- Indolent B-Cell (Experimental): Indolent B-Cell (IBCL): Small lymphocytic lymphoma, follicular lymphoma (Grade 1 or 2) and marginal zone lymphoma. Participants received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days
  Interventions: Drug: enzastaurin
- Aggressive B-Cell (Experimental): Aggressive B-Cell (ABCL): Primary central nervous system (CNS) lymphoma, follicular lymphoma (Grade 3a and 3b) and aggressive lymphoma with prior clinical history of indolent lymphoma. Participants received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days
  Interventions: Drug: enzastaurin

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose then 500 mg, oral, daily until progressive disease
  Other Names: LY317615

SUMMARY:
In this study, all patients will get investigational drug. There will be no comparator drug. This study will evaluate three tumor types: T-cell lymphoma, Indolent B-cell lymphoma, and Aggressive B-cell lymphoma. Each tumor type will include several tumor subtypes:

* T-cell lymphoma: Peripheral and Cutaneous T-cell lymphoma (PTCL, CTCL)
* Indolent B-cell lymphoma: Small lymphocytic lymphoma, follicular lymphoma (Gr 1 or 2) and marginal zone lymphoma
* Aggressive B-cell lymphoma: Primary CNS lymphoma, follicular lymphoma (Gr 3a and 3b) and aggressive lymphoma with prior clinical history of indolent lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Have measurable lesions
* Have recovered from prior chemotherapies
* Have an estimated life expectancy of at least 12 weeks
* Hepatic: total bilirubin less than or equal to 1.5 XULN; ATL/AST less than or equal to 2.0 x ULN (less than 5x if liver metastases are present)
* Renal: serum creatinine less than or equal to 1.5XULN
* Adequate bone marrow reserve: platelets greater than or equal to 75 x 109 /Liter (L) Criteria:
* Have a second primary malignancy (except adequately treated nonmelanomatous skin cancer, or other cancer that is considered cured by surgical resection or radiation).
* Anti-lymphoma therapy within the past 3 weeks
* Unable to swallow tablets
* Unable to discontinue use of carbamazepine, phenobarbital and phenytoin at least 14 days prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California, United States
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garran, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gosford, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auchenflower, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prahran, Victoria
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasília
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaú
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tepic
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalpan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Forsyth CJ, Gomez-Almaguer D, Camargo JF, Eliadis PE, Crespo-Solis E, Pereira J, Gutierrez-Aguirre CH, Rivas-Vera S, Roberson S, Lin B, Smith NV, Hamid O. A multicenter, open-label, noncomparative screening study of enzastaurin in adult patients with non-Hodgkin lymphomas. Clin Lymphoma Myeloma Leuk. 2013 Aug;13(4):398-403. doi: 10.1016/j.clml.2013.03.005. Epub 2013 Jun 14. PMID 23770158
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who had progressive disease, died due to any cause or alive and on study at the end of study, but off treatment.
Groups:
- T-Cell (TCL): T-Cell (TCL): Peripheral and cutaneous T-cell lymphoma (PTCL, CTCL). Participants received enzastaurin 1125 milligram (mg) loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Indolent B-Cell (IBCL): Indolent B-Cell (IBCL): Small lymphocytic lymphoma, follicular lymphoma (Grade 1 or 2) and marginal zone lymphoma. Participants received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Aggressive B-Cell (ABCL): Aggressive B-Cell (ABCL): Primary central nervous system (CNS) lymphoma, follicular lymphoma (Grade 3a and 3b) and aggressive lymphoma with prior clinical history of indolent lymphoma. Participants received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
Period: Overall Study
Arm/Group | T-Cell (TCL) | Indolent B-Cell (IBCL) | Aggressive B-Cell (ABCL)
Started | 23 | 19 | 15
Received At Least One Dose of Study Drug | 23 | 19 | 15
Progressive Disease | 15 | 11 | 7
Death | 1 | 1 | 2
Completed | 16 | 12 | 9
Not Completed | 7 | 7 | 6
Not completed — Adverse Event | 1 | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Physician Decision | 2 | 2 | 1
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- T-Cell: T-Cell (TCL): Peripheral and cutaneous T-cell lymphoma (PTCL, CTCL). Participants received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Total: Total of all reporting groups
Arm/Group | T-Cell | Indolent B-Cell | Aggressive B-Cell | Total
Number analyzed (Participants) | 23 | 19 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (17.54) | 69.7 (10.46) | 60.1 (8.44) | 58.9 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 7 | 24
  Male | 11 | 14 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 8 | 11 | 37
  Not Hispanic or Latino | 5 | 11 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 0 | 0 | 2
  White | 9 | 17 | 12 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 2 | 2 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 1 | 3
  Brazil | 7 | 2 | 3 | 12
  Mexico | 9 | 6 | 7 | 22
  Australia | 1 | 9 | 2 | 12
  Peru | 5 | 0 | 0 | 5
  Argentina | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (RR) (Percentage of Participants Exhibiting Complete Response [CR] or Complete Response Unconfirmed [CRu] or Partial Response [PR])
Description: Tumor RR is defined as the number of responders divided by the number of treated participants for that tumor subtype. A responder was a participant who exhibited: a CR defined as a modified severity-weighted assessment tool (mSWAT) value of zero or a partial response (PR) defined as a mSWAT value > 50% decrease from baseline [for participants with cutaneous T-cell lymphoma (CTCL) using the mSWAT or CR, unconfirmed CR (Cru), or PR as defined by Abrey et al., (2005) (for participants with central nervous system (CNS) Lymphoma); or for all other participants a CR or complete response - unconfirmed (CRu) or PR as defined by Cheson et al., (1999).
Time Frame: Baseline to Measured Progressive Disease (Up to 114 Months)
Population: All participants with all tumor subtypes, who received at least one dose of study drug, and had evaluable tumor response rate data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Peripheral T-cell Lymphoma (PTCL): Participants who had PTCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Cutaneous T-cell Lymphoma (CTCL): Participants who had CTCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Small Lymphocytic Indolent B-Cell Lymphoma (IBCL): Participants who had small lymphocytic IBCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Follicular Grade 1 & 2 (IBCL): Participants who had follicular grade 1 & 2 IBCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Marginal Zone Lymphoma (IBCL): Participants who had marginal zone lymphoma IBCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Follicular Grade 3a & 3b Aggressive B-cell Lymphoma (ABCL): Participants who had follicular grade 3 a ABCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- History of IBCL (ABCL): Participants who had a history of IBCL (ABCL) tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
Arm/Group | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Small Lymphocytic Indolent B-Cell Lymphoma (IBCL) | Follicular Grade 1 & 2 (IBCL) | Marginal Zone Lymphoma (IBCL) | Follicular Grade 3a & 3b Aggressive B-cell Lymphoma (ABCL) | History of IBCL (ABCL)
Number analyzed (Participants) | 12 | 11 | 7 | 8 | 4 | 5 | 10
percentage of participants
  CR | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 10.0 [0.3 to 44.5]
  CRu | 0 [0 to 0] | 9.1 [0.2 to 41.3] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  PR | 0 [0 to 0] | 9.1 [0.2 to 41.3] | 14.3 [0.4 to 57.9] | 12.5 [0.3 to 52.7] | 0 [0 to 0] | 20.0 [0.5 to 71.6] | 0 [0 to 0]
  Stable Disease | 33.3 [9.9 to 65.1] | 36.4 [10.9 to 69.2] | 85.7 [42.1 to 99.6] | 62.5 [24.5 to 91.5] | 100.0 [39.8 to 100] | 20.0 [0.5 to 71.6] | 50.0 [18.7 to 81.3]
  Progressive Disease (PD) | 50.0 [21.1 to 78.9] | 36.4 [10.9 to 69.2] | 0 [0 to 0] | 12.5 [0.3 to 52.7] | 0 [0 to 0] | 40.0 [5.3 to 85.3] | 30.0 [6.7 to 65.2]
  Unknown | 16.7 [2.1 to 48.4] | 9.1 [0.2 to 41.3] | 0 [0 to 0] | 12.5 [0.3 to 52.7] | 0 [0 to 0] | 20.0 [0.5 to 71.6] | 10.0 [0.3 to 44.5]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of study enrollment to the first date of objectively determined progressive disease or death from any cause. Progressive disease (PD) is an increase of Sézary cell percentage by greater than or equal to 40% in cluster of differentiation (CD4+/CD7- or 30% in CD4+/CD26- as compared to each respective nadir. mSWAT, primary central nervous system lymphoma (PCSNSL) and International Workshop Response Criteria (IWRC) response criteria were used for CTCL, primary central nervous system lymphoma (CNSL) and all other participants respectively. PFS was censored at the date of the last objective progression-free assessment.
Time Frame: Baseline to Measured Progressive Disease or Death From Any Cause (Up to 114 Months)
Population: All participants with all tumor subtypes, who received at least one dose of study drug and had evaluable PFS data. Participants censored: 0 (PTCL), 3 (CTCL), 0 (small lymphocytic), 2 (follicular grade 1 & 2), 0 (follicular grade 3a and 4b), 0 (marginal zone) and 4 (history of IBCL)
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- PTCL: Participants who had PTCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- CTCL: Participants who had CTCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Small Lymphocytic (IBCL): Participants who had small lymphocytic IBCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- Follicular Grade 3a & 4b (ABCL): Participants who had follicular grade 3 & 4 ABCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- History of IBCL (ABCL): Participants who had history of IBCL (ABCL) tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
Arm/Group | PTCL | CTCL | Small Lymphocytic (IBCL) | Follicular Grade 1 & 2 (IBCL) | Marginal Zone Lymphoma (IBCL) | Follicular Grade 3a & 4b (ABCL) | History of IBCL (ABCL)
Number analyzed (Participants) | 12 | 11 | 7 | 8 | 4 | 5 | 10
Days | 58 [23 to 95] | 227 [31 to 761] | 303 [113 to 342] | 429 [51 to 672] | 159 [67 to 168] | 114 [27 to 547] | 68 [11 to NA] — The upper limit could not be calculated due to the small number of events.

3. Secondary Outcome: Time to Progressive (TTP) Disease
Description: TTP disease is defined as the time from the date of study enrollment to the date of objectively determined disease progression. Objectively determined progressive disease (PD) was interpreted as meeting the criteria for PD. For patients who died without documented objective PD (including death from study disease); TTP was censored at the date of the last objective progression-free disease assessment prior to death. For participants not known to have died as of the data cut-off date and who did not have objective PD, TTP was censored at the date of the last objective progression-free disease assessment. For participants who received subsequent anticancer therapy (after discontinuation from study treatment) prior to objectively determined disease progression, TTP was censored at the date of the last objective progression free disease assessment prior to post-discontinuation therapy.
Time Frame: Baseline to Measured Progressive Disease (Up to 114 Months)
Population: All participants with all tumor subtypes, who received at least one dose of study drug and had evaluable TTP data. Participants censored: 0 (PTCL), 3 (CTCL), 0 (small lymphocytic), 2 (follicular grade 1 & 2), 0 (follicular grade 3a and 4b), 0 (marginal zone) and 4 (history of IBCL)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PTCL | CTCL | Small Lymphocytic (IBCL) | Follicular Grade 1 & 2 (IBCL) | Marginal Zone Lymphoma (IBCL) | Follicular Grade 3a & 4b (ABCL) | History of IBCL (ABCL)
Number analyzed (Participants) | 12 | 11 | 7 | 8 | 4 | 5 | 10
Days | 58 [23 to 95] | 227 [31 to 761] | 308 [113 to 556] | 429 [51 to 672] | 159 [67 to 168] | 114 [27 to 547] | 68 [11 to NA] — The upper limit could not be calculated due to the small number of events.

4. Secondary Outcome: Duration of Response (DOR)
Description: DoR is defined as the time from the date when the measurement criteria were met for CR, CRu, or PR (whichever status was recorded first) until the date of first observation of objectively determined disease progression (CR, CRu, or PR see above definition of responder). For responding participants who died without PD (including death from study disease), DoR was censored at the last assessment demonstrating lack of progression. For responding patients not known to have died as of the data cut-off date and who did not have PD, DoR was censored at the last assessment demonstrating objective response prior to the data cut-off date. For responding participants who received subsequent anticancer therapy (after discontinuation from the study treatment) prior to disease progression, DoR was censored at the last assessment demonstrating objective response prior to the initiation of post-discontinuation anticancer therapy.
Time Frame: Baseline to Measured Progressive Disease (Up to 97 Months)
Population: All participants with all tumor subtypes, who received at least one dose of study drug and had evaluable DOR data.
Measure: Median (Full Range); unit: Days
Groups:
- Marginal Zone Lymphoma Disease (IBCL): Participants who had marginal zone lymphoma (IBCL) tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
Arm/Group | PTCL | CTCL | Small Lymphocytic (IBCL) | Follicular Grade 1 & 2 (IBCL) | Marginal Zone Lymphoma Disease (IBCL) | Follicular Grade 3a & 4b (ABCL) | History of IBCL (ABCL)
Number analyzed (Participants) | 12 | 11 | 7 | 8 | 4 | 5 | 10
Days | 0 [0 to 0] | 394.0 [141.0 to 647.0] | 281.0 [281.0 to 281.0] | 1.0 [1.0 to 1.0] | 0 [0 to 0] | 58.0 [58.0 to 58.0] | 2957.0 [2957.0 to 2957.0]

5. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 1-Year
Description: PFS at 1 year was defined as the probability of being alive and having not progressed at 1 year and calculated from the PFS Kaplan-Meier analysis. PFS was censored at the date of the last objective progression-free assessment. Progressive disease (PD) is an increase of Sézary cell percentage by greater than or equal to 40% in cluster of differentiation (CD4+/CD7- or 30% in CD4+/CD26- as compared to each respective nadir. mSWAT, primary central nervous system lymphoma (PCSNSL) and International Workshop Response Criteria (IWRC) response criteria were used for CTCL, primary central nervous system lymphoma (CNSL) and all other participants respectively. PFS was censored at the date of the last objective progression-free assessment.
Time Frame: Baseline to Measured Progressive Disease or Death From Any Cause (1 Year)
Population: All participants with all tumor subtypes, who received at least one dose of study drug and had evaluable 1-year rate PFS data.
Measure: Number; unit: percentage of participants
Groups:
- Follicular Grade 3 & 4 (ABCL): Participants who had follicular grade 3 & 4 ABCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
- History of IBCL (ABCL): Participants who had history of IBCL ABCL tumor subtype and received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
Arm/Group | PTCL | CTCL | Small Lymphocytic (IBCL) | Follicular Grade 1 & 2 (IBCL) | Marginal Zone Lymphoma Disease (IBCL) | Follicular Grade 3 & 4 (ABCL) | History of IBCL (ABCL)
Number analyzed (Participants) | 12 | 11 | 7 | 8 | 4 | 5 | 10
percentage of participants | 0.0 | 36.8 | 14.3 | 51.4 | 0.0 | 25.0 | 48.6

6. Secondary Outcome: Number of Participants With One or More Drug-Related Adverse Events
Description: Number of participants with one or more Drug-Related Adverse Events. Clinically significant events are defined as serious adverse events, regardless of causality. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline to End of Study (Up to 114 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- T-Cell; Indolent B-Cell; Aggressive B-Cell: Participants received enzastaurin 1125 mg loading dose then 500 mg, oral, daily until progressive disease or predefined criteria for discontinuation is met. Participants who progress within the first 28 days may remain on study treatment, provided that the participant is not in need of immediate treatment with another anticancer therapy. Study treatment occurs in cycles. 1 cycle = 28 days.
Arm/Group | T-Cell | Indolent B-Cell | Aggressive B-Cell
Number analyzed (Participants) | 23 | 19 | 15
Participants | 2 | 3 | 0

ADVERSE EVENTS:
Time Frame: Up to 114 months
Description: Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly
Arm/Group | T-Cell | Indolent B-Cell | Aggressive B-Cell
Serious Adverse Events (participants affected / at risk) | 9/23 | 11/19 | 5/15
Other Adverse Events (participants affected / at risk) | 19/23 | 17/19 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Cell (N=23) | Indolent B-Cell (N=19) | Aggressive B-Cell (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 4 (5) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | T-Cell (N=23) | Indolent B-Cell (N=19) | Aggressive B-Cell (N=15)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 3 (11) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 2 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (4)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Vestibular neuronitis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (14) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Gingival erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (3)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 7 (10) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oedema (General disorders) | 0 (0) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 3 (4) | 3 (6)
Pyrexia (General disorders) | 6 (8) | 3 (3) | 1 (4)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood urea decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 3 (6) | 4 (5) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (4) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 1/11 (3) | 0/14 (0) | 0/8 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/11 (2) | 1/14 (1) | 0/8 (0)
Genital discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0/11 (0) | 1/14 (1) | 0/8 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/12 (0) | 0/5 (0) | 1/7 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1/11 (2) | 0/14 (0) | 0/8 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (5) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days